CLINICAL TRIAL: NCT03437018
Title: COMPARISON OF MONITORING OF MODERATE DIABETIC RETINOPATHY BY TELE-EXPERTISE AND CONVENTIONAL OPHTHALMOLOGICAL CONSULTATION
Brief Title: MONITORING OF MODERATE DIABETIC RETINOPATHY BY TELE-EXPERTISE
Acronym: TELERETINODIAB
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: ID RCB 2017-A02329-44
Record Dates: First submitted 2018-01-26; First posted 2018-02-19 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Diabetic Retinopathy
Keywords: moderate diabetic retinopathy; tele-expertise
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: moderate diabetic retinopathy follow-up by tele-expertise — Consultation by an orthoptist to measure visual acuity, eye tone by pulsed air tonometer, and retinography images after pupillary dilatation (9 photographs: one of the posterior pole and 8 of the peripheral retina) and optical coherence tomography (OCT).
  The results are immediately evaluated on site by an ophthalmologist. The results are sent through a secure online medical application to a diabetic retinopathy specialist ophthalmologist for evaluation.

SUMMARY:
The aim of this study is to evaluate the monitoring of moderate diabetic retinopathy by tele-expertise

DETAILED DESCRIPTION:
This study compares 2 strategies of monitoring of moderate diabetic retinopathy (RD).After a consultation with an orthoptist for measurement of visual acuity, measurement of ocular tone by pulsed air tonometer, retinography pictures (9 photographs: one of the posterior pole and 8 of the retinal periphery) and Optical Coherence Tomography (OCT), results are evaluated on-site by an ophthalmologist and then sent through a secure medical online application to an ophthalmologist expert in RD for assessment. Each patient is his own control.

ELIGIBILITY:
Inclusion Criteria:

* patient with complicated diabetes mellitus with moderate retinopathy

Exclusion Criteria:

* Patient deprived of liberty by judicial or administrative decision
* Person subject to a legal protection measure
* Patient already involved in another clinical trial protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with complicated diabetes mellitus with moderate retinopathy requiring periodic follow-up by an ophthalmologist
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
classification of diabetic retinopathy (DR) | 1 month
  DR is classified in 3 stages : moderate non proliferative DR, severe non proliferative DR, and proliferative DR

SECONDARY OUTCOMES:
classification of macular edema | 1 month
  macular edema (ME) is classified in 4 stages : no ME , mild ME, moderate ME, severe ME
follow-up strategy | 1 month
  follow-up strategy can take to ways : no treatment required and continuation of the monitoring/ complementary exam or treatment required
medical time necessary for examination and analyse | 1 month
  time necessary for direct examination and analyse by ophthalmologist on-site and time necessary for remote analyse are measured

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Penfornis, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schulze-Dobold C, Erginay A, Robert N, Chabouis A, Massin P. Ophdiat((R)): five-year experience of a telemedical screening programme for diabetic retinopathy in Paris and the surrounding area. Diabetes Metab. 2012 Nov;38(5):450-7. doi: 10.1016/j.diabet.2012.05.003. Epub 2012 Jul 4. PMID 22765981
- [Background] Chabouis A, Berdugo M, Meas T, Erginay A, Laloi-Michelin M, Jouis V, Guillausseau PJ, M'bemba J, Chaine G, Slama G, Cohen R, Reach G, Marre M, Chanson P, Vicaut E, Massin P. Benefits of Ophdiat, a telemedical network to screen for diabetic retinopathy: a retrospective study in five reference hospital centres. Diabetes Metab. 2009 Jun;35(3):228-32. doi: 10.1016/j.diabet.2008.12.001. Epub 2009 Apr 5. PMID 19349202
- [Background] Erginay A, Chabouis A, Viens-Bitker C, Robert N, Lecleire-Collet A, Massin P. OPHDIAT: quality-assurance programme plan and performance of the network. Diabetes Metab. 2008 Jun;34(3):235-42. doi: 10.1016/j.diabet.2008.01.004. PMID 18424210